CLINICAL TRIAL: NCT03717857
Title: A Sleep Hygiene Intervention to Improve Sleep Quality in Urban, Latino Middle School Children - Phase 1
Status: Completed | Type: Observational
Sponsor: Rhode Island Hospital (Other)
Collaborators: University of Puerto Rico (Other)
Responsible Party: Sponsor
Other Study IDs: 1R34HL135073 -Phase1; 1R34HL135073 (NIH)
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Sleep; Sleep Hygiene, Inadequate
Keywords: Latino children; middles school; sleep hygiene; educational intervention
MeSH Terms: conditions — Sleep Hygiene

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Caregiver InDepth Interviews: Caregivers who have a child between the ages of 11-13, who attends 6th-8th grades in one the targeted schools, and who resides in one of the targeted public school districts identified by zip code. In RI , caregivers will identity as Latino . Caregivers will participate in a one time in-depth qualitative interview regarding their child's sleep.
- Focus Groups: Three focus groups with middle school students [N = 5], caregivers [N =5], and school staff [N = 5] will be conducted to inform the development of the intervention.
  Criteria for caregiver and middle school student selection is similar to the in-depth interviews and the pilot clinical trial. Inclusion criteria specify that participants must 1) be between the ages of 11-13 , 2) be in 6th-8th grades, or have a child that meets that criteria 3) reside in one of the targeted public school districts identified by zip code, 4) attend one of the schools within these districts.In RI, caregivers will have to identify as Latino.
  The school staff focus group will include school personnel from the targeted schools.

SUMMARY:
Sleep is essential for children's daytime functioning and health. Poorer sleep hygiene can negatively affect sleep outcomes in children. Urban Latino children are at greater risk for poor sleep hygiene and poor quality sleep due to exposure to higher levels of urban and cultural stressors. This project aims to refine and test a novel school-based intervention to improve sleep hygiene and in turn, sleep quality in urban Latino middle school children. An existing sleep hygiene intervention that has been shown to improve sleep in urban children will be culturally and contextually tailored and has the potential to exert greater improvements in sleep hygiene and sleep outcomes for this high-risk group.

DETAILED DESCRIPTION:
Not sleeping long or soundly enough can lead to health problems in children, including more asthma symptoms and risk for obesity. Latino children might be especially at risk for poor sleep and worse asthma. Therefore, the goal of this study is to adapt an existing intervention called Sleep Smart for use with urban Latino middle school students. The new program will be called "Sleep Smart Latino" (SSL), the goal of which is to improve sleep quality among Latino, middle school-aged children in urban public schools. SSL will be administered by trained community members to a group of Latino middle school children who are at risk for poor sleep quality. The program will be tested in San Juan, Puerto Rico and Providence, Rhode Island.

The first aim of this project is to refine the SS intervention and intervention procedures so that they eventually can be used in a larger study of the intervention's effectiveness. Refinement will involve a) translation and cultural tailoring for Latino middle school students, b) enhancement of the parent component, and c) ensuring applicability to the urban, middle school setting in both sites (PR and RI). In-depth interviews with caregivers (N=20-25), focus groups (middle school students [N = 5], caregivers [N =5], and school staff [N = 5]), and Investigators with expertise in culturally tailored interventions will provide input.

The second aim of this project is to test the feasibility of the SSL intervention and training procedures through an Open Trial, to refine intervention modules and the training approach that will be used in the larger study. The Open Trial will include 15 adolescent participants at each study site.

The third aim of this project is to test the SSL intervention through a Pilot Randomized Control Trial (RCT) to provide estimates of effect size that will be used to inform the sample size for the larger study. The RCT will include 75 adolescent participants at each study site. We expect the participants in the SSL intervention will have improvement on the following primary sleep quality outcomes (improved sleep duration and sleep efficiency) as measured by actigraphy, relative to the control conditions. Secondarily, we expect participants in SSL will show a decrease in total daily caloric intake relative to the control conditions.

This registration refers only to aim 1 of the project.

ELIGIBILITY:
Inclusion Criteria:

* specify that participants must

  1. Be between the ages of 11-13,
  2. Be in 6th-8th grades,
  3. Reside in one of the targeted public school districts identified by zip code,
  4. Attend one of the schools within these districts,

Exclusion Criteria:

- 1) significant developmental delay, and/or severe psychiatric or chronic medical condition that preclude completion of study procedures or confound analyses.

2) current/prior sleep disorder diagnosis, such as sleep disordered breathing, restless leg syndrome, or periodic limb movement disorder (PLMD)

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population is urban, Latino middle school students (11-13 years old) and their primary caregivers. While for the second phase of this study participants will be middle school students who report sleeping less than 9 hours per night, for this phase those who sleep more and less than 9 hours per night will be included.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
cultural beliefs related to sleep behaviors and sleep health | Assessed one time ( 1 day at in -depth interview or focus group)
  Open ended questions that will examine cultural beliefs related to sleep behaviors, and sleep health, barriers to optimal sleep hygiene behaviors and strategies to ensure good sleep health
content and feasibility of the intervention | Assessed one time ( 1 day at in -depth interview or focus group)
  Open ended question will assess the helpfulness of key intervention components and strategies to engage students and to ensure caregiver involvement in the intervention.
Barriers and facilitators of intervention implementation in schools | Assessed one time ( 1 day school personnel focus group)
  Open ended question will solicit feedback on project barriers, resources and logistics to implementation within a school setting.

CONTACTS AND LOCATIONS:
Overall Officials: Daphne T Koinis-Mitchell, PhD, Principal Investigator — RI Hospital; Glorisa Canino, PhD, Principal Investigator — University of Puerto Rico
Locations (2):
- Rhode Island Hospital, Providence, Rhode Island, United States
- University of Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No